CLINICAL TRIAL: NCT00309569
Title: A Randomized Phase III Study Comparing Pre- and Postoperative vs. Conventional Adjuvant Treatment Hormone Receptor-negative Breast Cancer Patients
Brief Title: Randomized Study Comparing Pre- and Postoperative vs. Conventional Adjuvant Treatment in Receptor-negative Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Austrian Breast & Colorectal Cancer Study Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABCSG-7
Record Dates: First submitted 2006-03-31; First posted 2006-04-03 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Early Stage Breast Cancer
Keywords: Cyclophosphamide; Methotrexate; Fluorouracil; Epirubicine; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Methotrexate; Fluorouracil; Epirubicin; Surgical Procedures, Operative

ARMS (2):
- A (pre- + postoperative chemotherapy) (Experimental): 3 cycles CMF (cyclophophamide + Methotrexat + 5-Fluorouracil) followed by surgery. Subsequently node-positive patients received 3 cycles anthracycline-based chemotherapy regime EC (epirubicin + cyclophosphamide) and node-negative patients another 3 cycles CMF.
  Interventions: Drug: Cyclophosphamide; Drug: Methotrexate; Drug: Fluorouracil; Drug: Epirubicin; Other: Surgery
- B (conventional postoperative chemotherapy) (Experimental): Surgery followed by 3 cycles CMF (cyclophophamide + Methotrexat + 5-Fluorouracil). Subsequently node-positive patients received 3 cycles anthracycline-based chemotherapy regime EC (epirubicin + cyclophosphamide) and node-negative patients another 3 cycles CMF.
  Interventions: Drug: Cyclophosphamide; Drug: Methotrexate; Drug: Fluorouracil; Drug: Epirubicin; Other: Surgery

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide 600mg/m2
Drug: Methotrexate — Methotrexate 40mg/m2
Drug: Fluorouracil — Fluorouracil 600mg/m2
Drug: Epirubicin — Epirubucin 60mg/m2 (only node-positive patients)
Other: Surgery — Surgery

SUMMARY:
Primarily, this clinical investigation compared overall survival and recurrence-free survival in patients with hormone receptor-negative breast cancer treated with pre- and postoperative chemotherapy vs. conventional postoperative treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with bioptically verified breast cancer
* Estrogen receptor-negative status
* Age: < 70 years
* WHO Performance Status < 2
* Laboratory parameters

  1. hematopoiesis: > 3500/mm3 leukocytes, > 100,000/mm3 thrombocytes
  2. renal function: creatinin < 1.5mg%
  3. hepatic function: GOT max. 2.5 x UNL
  4. bilirubin: < 2.0 mg %
  5. metabolic parameters: Na, Ca, K in normal range
* </= 4 weeks interval since surgery
* Informed consent

Exclusion Criteria:

* Patients with locally inoperable cancer, M1
* Other preoperative tumor-specific radiotherapy, chemotherapy or endocrine treatment
* Pregnancy or lactation
* General contraindication against cytostatic treatment
* T4 cancer; inflammatory disease, simultaneous or sequential bilateral breast cancer
* Lacking compliance or understanding of disease
* Serious concomitant disease
* Second carcinoma or status post second carcinoma (except for treated squamous cell carcinoma of the skin or cervical carcinoma in situ)

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 429 (Actual)
Dates: Start 1991-10 (Actual); Primary Completion 2000-09 (Actual); Study Completion 2000-09 (Actual)

PRIMARY OUTCOMES:
Overall survival
Recurrence-free survival

SECONDARY OUTCOMES:
Rate of breast-conserving procedures

CONTACTS AND LOCATIONS:
Overall Officials: Raimund Jakesz, MD, Principal Investigator — Austrian Breast & Colorectal Cancer Study Group

REFERENCES:
- See also: Related Info — http://www.abcsg.at